CLINICAL TRIAL: NCT00038701
Title: Phase II Study of Gemcitabine-Based Chemoradiation and TNP-470 for Patients With Locally Advanced, Nonmetastatic Adenocarcinoma of the Pancreas
Brief Title: Study of Gemcitabine Chemoradiation and TNP-470 Patients Locally Advanced, Nonmetastatic Adenocarcinoma of Pancreas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID98-248
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Metastatic Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — O-(Chloroacetylcarbamoyl)fumagillol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemzar Chemoradiation + TNP-470 (Experimental)
  Interventions: Drug: TNP-470

INTERVENTIONS:
Drug: TNP-470

SUMMARY:
The goal is to assess survival and patterns of failure in patients treated with Gemzar-based chemoradiation and TNP-470 for locally advanced adenocarcinoma of the pancreas.

ELIGIBILITY:
Patients must have cytologic or histologic proof of adenocarcinoma of the pancreas.

All patients must be staged with a physical exam and CXR. Patients must have locally advanced disease defined as tumor extension to the celiac axis or SMA, or occlusion of the SMPV confluence (on contrast-enhanced CT). There must be no radiographic evidence of metastatic disease.

Patients must have had no prior chemotherapy or irradiation.

Patients must have a baseline Karnofsky performance status of at least 60.

Patients must have adequate bone marrow reserve platelet count >100,000/mL, hemoglobin>9 g/dL, absolute granulocyte count must be >1,500 cells/mm3,serum creatinine must be <1.6 mg/dL. Serum bilirubin must be less than 5 mg/dL prior to therapy with endoscopic or percutaneous drainage if necessary.

Patients must have estimated life expectancy of at least 12 weeks.

Patients must be at least 18 years of age. There will be no upper age restriction.

Female patients must have had childbearing potential terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, barrier device, or abstinence.

Patients cannot have hepatic or peritoneal metastases detected by ultrasound (US), CT scan, or laparotomy prior to chemoradiation.

Before receiving external beam irradiation, patients should be able to maintain adequate oral nutrition (90% to 100% of estimated need of calories and protein) and be free of significant nausea and vomiting.

Patients should have bilateral renal function, as determined on excretory urogram (IVP) or abdominal CT, or >2/3 of one functioning kidney must be able to be shielded from the radiation beam.

Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude protocol therapy.

Patients must sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1999-08 (Actual); Primary Completion 2004-05-11 (Actual); Study Completion 2004-05-11 (Actual)

PRIMARY OUTCOMES:
Patient Survival Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B. Evans, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org